CLINICAL TRIAL: NCT06532786
Title: Neural Adaptations to Metronome-Paced Strength Training: Insights From Neuroscience and Human Movement Variability
Brief Title: Neural Adaptations to Metronome-Paced Strength Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: METROTRAIN - 1403
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Motor Control; Neuroscience; Neural Adapatations; Transcranial Magnetic Stimulation; Dynamic Systems; Metronome Paced Strength Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fractal Paced (Experimental): Strength training in single leg extension machine, synchronizing each repetition with a fractal-like visual metronome, i.e., a metronome presenting visual external cues with variability within its temporal structure.
  Interventions: Other: Fractal Paced
- Isochronous Paced (Experimental): Strength training in single leg extension machine, synchronizing each repetition with a isochronus visual metronome, i.e., a metronome presenting visual external cues withthe same pace in each repetition (without variability)
  Interventions: Other: Isochronous Paced
- Self Paced (Experimental): Strength training in single leg extension machine at participants self pace.
  Interventions: Other: Self Paced

INTERVENTIONS:
Other: Fractal Paced — The intervention consists in a metronome-paced strength training session performed 3 times per week (with 48h of rest between sessions), during 4 weeks. Each session consists in 4 sets of 15 repetitions at 65% of the one-repetition maximal (1RM) in single leg extension machine, synchronizing each repetition with fractal external cues presented by a visual metronome. The rest between sets will be set at 2 minutes of rest between sets.
  Arms: Fractal Paced
Other: Isochronous Paced — The intervention consists in a metronome-paced strength training session performed 3 times per week (with 48h of rest between sessions), during 4 weeks. Each session consists in 4 sets of 15 repetitions at 65% of the one-repetition maximal (1RM) single in leg extension machine, synchronizing each repetition with isochronus external cues presented by a visual metronome. The rest between sets will be set at 2 minutes of rest between sets.
  Arms: Isochronous Paced
Other: Self Paced — The intervention consists in a metronome-paced strength training session performed 3 times per week (with 48h of rest between sessions), during 4 weeks. Each session consists in 4 sets of 15 repetitions at 65% of the one-repetition maximal (1RM) in single leg extension machine, at their own self pace (with no metronome). The rest between sets will be set at 2 minutes of rest between sets.
  Arms: Self Paced

SUMMARY:
The aim of the study is to investigate the effects of incorporating variability within Resistance Training (RT) methods on the neural adaptations along the corticospinal tract and on neuromuscular function. The literature suggests that RTis one of the most common modalities to enhance and restore muscle function and its practice results in adaptation in neural and morphological adaptations. It is also known that conditions such as ageing and injury have a negative impact on neural drive to the muscles with consequences at motor control level that are not addressed by traditional RT. Recent approaches such as metronome paced strength training have been used to cover this motor control dimension through a greater control and consciousness of movement. However, this methodology tends not to incorporate the inherent variability and complex, fractal-like fluctuations that characterize human movement. The investigators propose that incorporating variability through a fractal-like metronome approach will speed up the neural adaptations which will be useful in injury rehab.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 40 years

Exclusion Criteria:

* Neurologic conditions;
* Lower limb disabilities or disease;
* Not able to provide informed consent;
* Have an implanted device (e.g. pacemakers) or any metal in the body;
* Medication advised against the application of Transcranial Magnetic Stimulation;
* History/family history of seizures, brain lesions or head trauma, neurological or psychiatric diseases, epilepsy, migraine

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Corticospinal Excitability (CSE) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  CSE is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of excitability of the corticospinal tract.
Short-interval Intracortical Inhibition (SICI) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  SICI is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of inhibition within the motor cortex.
Corticospinal Silent Period (CSP) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  CSP is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of inhibition along the corticospinal tract.
Intracortical Facilitation (ICF) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  ICF is a parameter extracted through the application of Transcranial Magnetic Stimulation (TMS). This parameter provides information regarding the level of facilitation within the motor cortex.
Lumbar Evoked Potentials (LEP) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  LEP is a measure extracted through the aplication of Lumbar stimulation. This measure allow to distinguish the adaptations that occur at spinal level as a result of strength training.
Maximal Compound Action Potentials (Mmax) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  Mmax is a measure assessed through peripheral nerve stimulation and represents the maximal capacity of recruit the motoneurons that innerve a muscle.
StartReact Gain changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  StartReact gain is a measure that is calculated following the StartReact protocol. It consists in measuring the participants' reaction times in response to visual stimuli (visual reaction time [VRT]), visual stimuli combined with a quiet sound (visual auditory reaction time [VART]) and visual startling stimuli (visual startling reaction time [VSRT]) and, then, apply the following formula: StartReact gain = ([VRT - VSRT]/[VRT - VART]).

SECONDARY OUTCOMES:
Single leg extension 1RM changes after 4-weeks intervention (PRE to POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  Single leg 1RM is defined as the maximal load that each participant mobilized in a single maximum dynamic knee extension.
Maximal Voluntary Isometric Contraction (MVIC) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  MVIC is defined as the maximal force an individual can produce against an immovable resistance
Sample Entropy (SampEn) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  SampEn is a non-linear measure of the temporal structure of force output, being an indicator of the regularity of this physiological output. It is obtained from sustained submaximal isometric contractions and it has been proposed as an indirect index of the capacity of the neuromuscular system to adapt the force output to changes in environment, i.e., its adaptability.
Coefficient ov variation (CV) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  CV is a common linear measure that translates the amount of variability within the signal and is calculated through the standard deviation normalised to the mean of a time series
Motor Unit Action Potentials (MUAP) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  MUAP is obtained through the decomposition of electromyographic (EMG) signals collected using High-density surface EMG electrodes and is an index of motor unit recruitment.
Firing Rate (FR) changes across the 4-weeks intervention (PRE to Week1, Week 2, Week 3, POST and follow-up) both within and between Fractal paced, Isochronus Paced and Self paced groups | PRE (baseline), W1 (week 1), W2 (week 2), W3 (week 3), POST (week 4), FUP (follow-up 4 weeks after the end of intervention)
  FR is obtained through the decomposition of electromyographic (EMG) signals collected using High-density surface EMG electrodes and is a measure of intramuscular coordination

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health & Science, Almada, Monte de Caparica, Portugal

IPD SHARING:
Plan to Share IPD: No